CLINICAL TRIAL: NCT05141812
Title: What is the Influence of Visual-motor Reliance on Planned and Unplanned Change of Direction Biomechanics 7 Months Post Anterior Cruciate Ligament Reconstruction?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sports Surgery Clinic, Santry, Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: SSC-ACL-003
Record Dates: First submitted 2021-11-03; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: ACL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACLR group: ACLR participants would be 7 months post surgery
- healthy control group: Healthy uninjured participants who are actively engaged in gaelic football or hurling.

SUMMARY:
The majority of anterior cruciate ligament (ACL) injuries occur during non-contact mechanisms.This suggests that an individual's movement technique is a significant factor in the cause of the injury. Hence, ACL injuries are increasingly being framed as an error in motor planning and execution.

Rehab following an ACL reconstruction (ACLR) commonly follows a pathway of: regaining ROM, strength development, power development, running, return to training and then return to competition. However, several studies utilising functional brain MRI and electroencephalogram have demonstrated dysfunction within the somatosensory and visual systems in the ACLR population even after the completion of rehabilitation. This has been suggested to indicate that the ACLR population becomes reliant on their visual system during motor planning and execution, potentially increasing the risk of reinjury.

DETAILED DESCRIPTION:
It has been demonstrated in studies utilising functional brain MRI and EEG that following ACLR, individuals have increased activation of the visual system during simple motor tasks as compared to healthy controls. This is suggested to represent an increased reliance on the visual system during motor planning and execution. Increased reliance on the visual system may negatively affect an individual's ability to respond to sporting situations which are often chaotic in nature, resulting in an inappropriate movement technique being employed. This may then result in an increased risk of reinjury. However, no study to date has been able to assess how visual reliance affects change of direction biomechanics.

The study will recruit individuals who are 7 months post-ACLR and intend on returning to multi-directional field sport. Individuals will complete a stepping down task (eyes open versus eyes closed) to identify participants who are reliant on their visual system. Participants will then complete a 90 deg change of direction task in a planned and then unplanned condition. Those who are visually reliant will be compared to those who are aren't with regards to their unplanned change of direction biomechanics and also the change in their biomechanics from a planned to unplanned condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years old
* Playing club level Gaelic football or hurling
* They must report that they intend on returning to sport at the same or higher level
* Able to give written informed consent and to participate fully in the interventions
* At 7 months biomechanical testing, individuals would need to have 70% symmetry of both quadriceps and hamstring peak torque as measured on our isokinetic dynamometer with the angular velocity set to 60°/s
* Individuals should have already commenced linear running and double leg jumping tasks as part of their rehabilitation
* They are currently attending a gym or can attain gym access for the duration of intervention period

Exclusion Criteria:

* They have not commenced running or jumping in their rehabilitation
* Revision ACL
* They underwent concurrent meniscal repair, chondral repair or extra-articular augmentation
* Serious medical conditions preventing them from completing high intensity resistance exercise
* Any previous: injuries to the visual system, concussion, head injury, unexplained seizures or epilepsy
* Any previous ankle or knee injuries
* Those who are uncomfortable or do not want to hop with their eyes closed (one of the assessment tasks will involve hopping on one leg with their eyes open and followed by another set in which their eyes are closed

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients would be recruited from those undergoing an ACLR under the care of orthopaedic surgeons at the Sports Surgery Clinic (Dublin, Ireland). At present, patients attend the Sports Medicine Department at Sports Surgery Clinic for strength, power and 3D biomechanical analysis at 7 months post-operatively prior to their reviews with their surgeon
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change of direction biomechanics- planned versus unplanned | at 7 months post-ACLR
  Participants will perform 90 degree cut within a 3D lab utilising using an eight-camera motion analysis system (200Hz: Bonita-B10, Vicon, UK) and integrated force plates (1000Hz BP400600, AMTI, USA). Timing gates (Smartspeed, Fusion Sport) will be used to time the change of direction and also provide the participant a visual stimulus as to which direction they need to cut to. The lights will be on during planned change of direction and 3 trials will be taken for each direction. During the unplanned change of direction, the target timing gates (right or left) will only switch on 2 metres prior to the participants approaching the force plates. 3 trials will be taken in the unplanned condition
Time to stability during stepdown task (eyes open versus eyes closed) | at 7 months post-ACLR
  Participants will stepdown from a 20cm box and land on one leg. Participants will be advised to achieve stability as quickly as possible and then to remain in that position for 20 seconds. Participants will complete 3 trials on each leg first with their eyes open and then a further 3 trials on each leg whilst blindfolded. Participants will perform this test in the 3D lab utilising using an eight-camera motion analysis system (200Hz: Bonita-B10, Vicon, UK)

SECONDARY OUTCOMES:
Joint position sense test | at 7 months post-ACLR
  Participants will be seated and blindfolded. Participants will perform this test in the 3D lab utilising using an eight-camera motion analysis system (200Hz: Bonita-B10, Vicon, UK). The assessor will active extend the participant's knee to between 0-30 degrees and hold it there. The participant will then be asked to replicate that angle 5 times for each leg
single leg balance (eyes open versus eyes closed) | at 7 months post-ACLR
  Participants will perform this test in the 3D lab utilising using an eight-camera motion analysis system (200Hz: Bonita-B10, Vicon, UK) and integrated force plates (1000Hz BP400600, AMTI, USA). Participants will stand on one leg with less than 15 degrees knee flexion. They will be asked to balance for 20 seconds. 3 trials will be taken for each leg with participants' eyes open and 3 trials of each leg whilst they are blindfolded
Quadriceps and hamstrings strength | at 7 months post-ACLR
  isokinetic dynamometry conducted on each leg between 0-100 degrees at 60 deg/sec. 3 sets of 5 completed for each leg
Countermovement jump- double and single leg | at 7 months post-ACLR
  Participants will be instructed to jump as high as they can. This will be conducted 3 times with double leg and then 3 trials single legged (for each leg)
Drop jump- double leg and single leg | at 7 months post-ACLR
  participants will drop off 30cm step (double leg) and 15cm step (single leg) and be instructed to quickly jump off the ground and as high as they can. 3 trials of each will be taken
anterior cruciate ligament return to sport after injury (ACL-RSI) questionnaire | at 7 months post-ACLR
  Questionnaire utilised to assess for participants' readiness to return to sport and identify if there are any potential psychological factors impacting their return to sport.
  Minimum score 0% and maximum score 100%. Lower score indicates less fear regarding return to sport
International knee documentation committee (IKDC) Questionnaire | at 7 months post-ACLR
  Questionnaire utilised to assess participants' self-reported function. Minimum score 0 and maximum score 100. A higher score indicates higher levels of function
Tampa scale of kinesiophobia | at 7 months post-ACLR
  Questionnaire utilised to assess participants' fear of movement or reinjury. Minimum score 17 and maximum score 68. A lower score indicates better outcome or reduced kinesiophobia
Near far quickness score (as part of visual processing software) | at 7 months post-ACLR
  sensory tablet (Senaptec, USA) with preloaded assessment tasks to across multiple visual processing domains including near far quickness task. The task requires the participants to correctly answer a task on a screen 3 metres away. Upon entry of the correct answer, a task appears on a device 70-100cm from the participant. The task will then continue to move between the 2 screens over a 30 second period, with the number of correct responses and time taken to input a response being calculated. The number of correct responses over 30 second test period is reported with a higher score indicating better function
Near far quickness reaction time to target (as part of visual processing software) | at 7 months post-ACLR
  sensory tablet (Senaptec, USA) with preloaded assessment tasks to across multiple visual processing domains including near far quickness task. The task requires the participants to correctly answer a task on a screen 3 metres away. Upon entry of the correct answer, a task appears on a device 70-100cm from the participant. The task will then continue to move between the 2 screens over a 30 second period, with the number of correct responses and time taken to input a response being calculated. Average response time is calculated for individual to input correct response for a far target and a near target. A lower value indicates quicker reaction time and hence better function.
Perception span (as part of visual processing software) | at 7 months post-ACLR
  sensory tablet (Senaptec, USA) with preloaded assessment tasks to across multiple visual processing domains including perception span task. The task involves recalling which circles were filled following a pattern being flashed for 1 second. Total score is calculated by the software with a higher score indicating better function
multiple object tracking score (as part of visual processing software) | at 7 months post-ACLR
  sensory tablet (Senaptec, USA) with preloaded assessment tasks to across multiple visual processing domains including multiple object tracking task. In the task, a set of circles are highlighted to the participant. The circles then spin around the screen in conjunction with other circles before coming to a stop. The participant is then tasked with correctly identifying the circles that were initially highlighted.The software provides a proportional and composite score. A higher score indicates better function
Reaction time (as part of visual processing software) | at 7 months post-ACLR
  sensory tablet (Senaptec, USA) with preloaded assessment tasks to across multiple visual processing domains including reaction time task. In the task, the participant places both index fingers on the screen, a flashing red image indicates which finger needs to be removed from the screen. The participant is advised to remove their finger from the screen as quickly as possible. Reaction times are provided by the software for each side (dominant hand and non-dominant hand) and also as an average between the two sides. A lower time indicates better function

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland